CLINICAL TRIAL: NCT02268708
Title: Evaluation of Post-operative Respiratory Complications After Thoracic Surgery in Patients With COPD
Status: Completed | Type: Observational
Sponsor: Hôpital Cochin (Other)
Responsible Party: Principal Investigator, Demiri Suela, Resident, Hôpital Cochin
Other Study IDs: COCHIN2014BPCO
Record Dates: First submitted 2014-08-06; First posted 2014-10-20 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: COPD; Malignant Neoplasm of Thorax
Keywords: COPD; Surgery, Thoracic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD: Patients:
  >18 years old COPD: FEV/FEV1<80% in respiratory evaluation who have un oncological pulmonary resection in Cochin Hospital Paris France
  Interventions: Procedure: Oncological pulmonary resection

INTERVENTIONS:
Procedure: Oncological pulmonary resection — Respiratory evaluation before sugery Oncological pulmonary resection with general anesthesia. Hospitalization for post operative care

SUMMARY:
Evaluation of post-operative respiratory complications after thoracic surgery for pulmonary resection in patients with COPD

Introduction: Postoperative pulmonary complications following pulmonary resection occur in 12-40% of cases. Some risk factors such as COPD are well identified. It has been shown that COPD patients with a history of frequent exacerbations are more likely to develop exacerbations. No study has evaluated the rate of patients called 'frequent exacerbators' among COPD patients requiring pulmonary resection and the relations between exacerbations history and incidence of acute respiratory postoperative complications.

The main objective is to determine the frequency of pulmonary postoperative complications (atelectasis, acute respiratory failure, pneumonia) following lung resection in COPD patients. The secondary objectives are to determine the frequency of extra pulmonary postoperative complications and the prevalence of the 'frequent exacerbator' phenotype in this population, as well as its relation with the risk of post-operative complications.

Materials and Methods: This is a prospective, observational, single-center study, of patients with COPD hospitalized for elective thoracic surgery in the center of Thoracic Surgery, Hôpital Cochin. The inclusion criteria are: male or female aged more than 40 years, permanent airflow obstruction as defined by an FEV/FVC ratio < 70% after bronchodilator. Collected data will be: COPD symptoms (dyspnea score, exacerbations) by a questionnaire given to the patient during the anesthesia consultation, COPD severity scores, comorbidities, per operative data, postoperative complications, hospitalization and intra-hospital mortality.

Perspectives: This work will provide information on the risk of postoperative complications in patients with COPD and the influence of the 'frequent exacerbator' phenotype. This will help adapting preventive care to the COPD subtype .

ELIGIBILITY:
Inclusion Criteria:

* Male or Female >40 years old
* COPD permanent airflow obstruction as defined by an FEV/FVC ratio < 70% after bronchodilator
* Hospitalized for elected surgical pulmonary resction

Exclusion Criteria:

* Pregnancy
* Patient under Long duration Oxygen
* Questionnaire information impossible to understand (because of language)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male or female aged more than 40 years, permanent airflow obstruction as defined by an FEV/FVC ratio < 70% after bronchodilator. Collected data will be: COPD symptoms (dyspnea score, exacerbations) by a questionnaire given to the patient during the anesthesia consultation, COPD severity scores, comorbidities, per operative data, postoperative complications, hospitalization and intra-hospital mortality.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of pulmonary postoperative complications lung resection in COPD patients. | 1 YEAR
  Evaluate the prevalence of atelectasis, acute respiratory failure and post operative pneumonia after thoracic surgery for lung resection in COPD (Chronic Obstructive Pulmonary Disease) patients.

SECONDARY OUTCOMES:
It is to determine the prevalence of the 'frequent exacerbator' phenotype in this COPD population, as well as its relation with the risk of post-operative complications. | 1 YEAR
Mortality | 30 days
Duration of total hospitalisation, and ICU hospitalisation | 30 days
Any other non respiratory complication | 30 days
  Coplications: cardiac, kiddney, sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Suela Demiri, Resident, Principal Investigator
Locations (1):
- Réanimation chirurgicale thoracique Hôpital Cochin, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Hurst JR, Vestbo J, Anzueto A, Locantore N, Mullerova H, Tal-Singer R, Miller B, Lomas DA, Agusti A, Macnee W, Calverley P, Rennard S, Wouters EF, Wedzicha JA; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Susceptibility to exacerbation in chronic obstructive pulmonary disease. N Engl J Med. 2010 Sep 16;363(12):1128-38. doi: 10.1056/NEJMoa0909883. PMID 20843247
- [Result] Wedzicha JA, Seemungal TA. COPD exacerbations: defining their cause and prevention. Lancet. 2007 Sep 1;370(9589):786-96. doi: 10.1016/S0140-6736(07)61382-8. PMID 17765528
- [Result] Wan ES, DeMeo DL, Hersh CP, Shapiro SD, Rosiello RA, Sama SR, Fuhlbrigge AL, Foreman MG, Silverman EK. Clinical predictors of frequent exacerbations in subjects with severe chronic obstructive pulmonary disease (COPD). Respir Med. 2011 Apr;105(4):588-94. doi: 10.1016/j.rmed.2010.11.015. Epub 2010 Dec 10. PMID 21145719